CLINICAL TRIAL: NCT05842252
Title: Single-stage Correction of Acute Angle Coxa Vara
Acronym: Coxavara
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hesham Mohamed Elbaseet, Dr., Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACUTECOXAVARA
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Coxa Vara
Keywords: coxa vara; proximal femur osteotomy; subtrochanteric valgus osteotomy; Wagner technique; tension band wiring.; greater trochanter transfer
MeSH Terms: conditions — Coxa Vara

STUDY DESIGN:
Intervention Model Description: greater trochanter transfer and subtrochanteric valgus osteotomy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- greater trochanter transfer and subtrochanteric valgus osteotomy (Experimental): greater trochanter transfer, subtrochanteric valgus osteotomy fixation by Wagner & TB and Locked plate
  Interventions: Procedure: greater trochanter transfer, subtrochanteric valgus osteotomy

INTERVENTIONS:
Procedure: greater trochanter transfer, subtrochanteric valgus osteotomy — greater trochanter transfer, subtrochanteric valgus osteotomy fixation by wagner TB and locked plate

SUMMARY:
Correction of sever degree of coxa vara in single-stage correction.

DETAILED DESCRIPTION:
The technique described in this article illustrates how to fully correct acute angle developmental coxa vara (neck shaft angle 30 degrees) to obtain better radiological and functional outcomes.

GT transfer Subtroch. valgus osteotomy

ELIGIBILITY:
Inclusion Criteria:

* acute coxa vara

Exclusion Criteria:

* osteopenic oI

Ages: 3 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
modified McKay's criteria | 1 year
  Hip function score
  1. Excelent
  2. Good
  3. Fair
  4. Poor

CONTACTS AND LOCATIONS:
Overall Officials: Hesaham M Elbaseet, MD, Principal Investigator — Assiut University
Locations (1):
- faculty of medicine Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Srisaarn T, Salang K, Klawson B, Vipulakorn K, Chalayon O, Eamsobhana P. Surgical correction of coxa vara: Evaluation of neck shaft angle, Hilgenreiner-epiphyseal angle for indication of recurrence. J Clin Orthop Trauma. 2019 May-Jun;10(3):593-598. doi: 10.1016/j.jcot.2018.06.009. Epub 2018 Jun 28. PMID 31061596
- [Background] Galal S. Percutaneous multiplanar subtrochanteric osteotomy with external fixation for developmental coxa vara (preliminary results). J Pediatr Orthop B. 2017 Jul;26(4):320-328. doi: 10.1097/BPB.0000000000000392. PMID 27748677